CLINICAL TRIAL: NCT06216899
Title: Reverse-Engineering of Exclusive Enteral Nutrition (RE-EEN) in Crohn's Disease: A Multi-Center Trial
Acronym: mRE-EEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Dale Lee, Associate Professor, Medical Director, Clinical Nutrition; Director of the Celiac Disease Program, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004459
Record Dates: First submitted 2024-01-04; First posted 2024-01-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
Keywords: Crohn's; Inflammatory Bowel Disease; CD
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smoothie (Experimental): In the smoothie arm, you will be provided instructions, a blender, and food components to prepare the smoothie at home.
  Interventions: Other: Whole-food based smoothie
- Formula (Active Comparator): In the formula arm, you will be given conventional formula as per the direction of the gastroenterology team along with our dieticians.
  Interventions: Other: Formula

INTERVENTIONS:
Other: Whole-food based smoothie — The smoothies will be based upon the concept of reverse-engineering of exclusive enteral nutrition and provide 100% of calculated caloric needs for weeks 0-4. At week 4, select foods will be introduced to provide up to 20% of daily caloric needs.
  Arms: Smoothie
Other: Formula — Conventional formula (Boost, Ensure, Modulen) as per the direction of their primary Gastroenterology team to provide 100% of calculated caloric needs for weeks 0-4. At week 4, select foods will be introduced to provide up to 20% of daily caloric needs.
  Arms: Formula

SUMMARY:
This study will compare the tolerability and efficacy of conventional formula Exclusive Enteral Nutrition (EEN) and whole-food blended smoothie EEN by enrolling a total of 60 participants with newly diagnosed pediatric Crohn's disease (CD).

Participants will be provided either commercial formula or guided on the preparation of the home-blended smoothie. These participants will be given a specific recipe, blender, and be provided the food components to the smoothie. The study will total 8 weeks and will assess tolerance, clinical outcomes, stool microbiome, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 -21 years old.
* Diagnosis of Crohn's disease within 24 months
* Elevation in objective inflammatory markers at enrollment: C-reactive protein (CRP), ESR, or fecal calprotectin
* Active Crohn's disease, as defined by Pediatric Crohn's Disease Activity Index (PCDAI) ≥10.
* Participant capable of giving informed consent, or if a minor the parent/guardian is capable of giving informed consent.

Exclusion Criteria:

* History of surgery for Crohn's disease.
* Perianal disease as part of Crohn's disease phenotype.
* Recent use of:
* corticosteroids (within 4 weeks),
* dose adjustment of immunomodulator (within 8 week)
* azathioprine 4 weeks prior to study final visit (week 8)
* start or adjust methotrexate 3 weeks prior to final study visit.
* Prior use of biological medication
* Prior treatment with EEN or other dietary therapy for Crohn's disease.
* Prior treatment with antibiotics for Crohn's disease.
* Known allergies to any of the food components in the smoothie.
* Admission to hospital due to severity of Crohn's disease and associated symptoms.
* Unwillingness to provide informed consent.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2030-01-10 (Estimated)

PRIMARY OUTCOMES:
Tolerance- Ability to remain on prescribed nutritional therapy | 4 and 8 weeks
  Tolerance of therapy as measured by ability to continue prescribed nutritional therapy over 4-weeks and 8-weeks without deviation from protocol. Participants will meet with a study dietitian at week 2, week4, and week 8. Dietitians will evaluate caloric needs, specific deficits, and dietary limitations.

SECONDARY OUTCOMES:
Fecal Calprotectin reduction from baseline | 4 and 8 weeks
  Fecal calprotectin (FCP) level <250 μg/gram
Pediatric Crohn's Disease Activity Index (PCDAI) reduction from baseline | 4 and 8 weeks
  Pediatric Crohn's Disease Activity Index (PCDAI) score <10 (clinical remission).
  PCDAI will be calculated at each visit. The total score is calculated from assessments in 11 sections. Minimum score 0. Maximum score 100. A lower score is better.
  History (recall 1 week)
  * Abdominal pain
  * Stools
  * Patient functioning
  * General well-being
  Physical Examination
  * Weight
  * Height
  * Abdomen
  * Peri-rectal disease
  * Extra-intestinal manifestations
  Laboratory
  * Hematocrit (%)
  * Erythrocyte sedimentation rate (ESR) (mm/hr)
  * Albumin (g/L)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Lee, MD, MSCE, Principal Investigator — Seattle Children's Hospital, University of Washington
Locations (3):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Izaak Walton Killam Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No